CLINICAL TRIAL: NCT01846000
Title: Evaluation of Effect of Low-level Laser Therapy on Adolescents With Temporomandibular Disorder
Brief Title: Low-level Laser Therapy on Temporomandibular Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Camila Haddad Leal de Godoy, Master Student, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLLTMD 40455
Record Dates: First submitted 2013-04-11; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Temporomandibular Disorder
Keywords: temporomandibular joint; temporomandibular disorder; electromyography; low-level laser therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Muscles of mastication (Experimental): This group with TMD will receive low-level laser treatment at masseter and temporal muscles - three points on the masseter (upper, middle and lower) and one point on the anterior temporal
  Interventions: Procedure: low-level laser treatment
- TMJ and muscles (Experimental): This group with TMD will receive a mixed application of low-level laser treatment- TMJ and muscles of mastication.
  Interventions: Procedure: low-level laser treatment
- Placebo (Placebo Comparator): This group with TMD will receive a low-level laser placebo treatment at TMJ and muscles of mastication. The same equipment will be used with a pen that emits a red guide light and a warning sound, but without the emission of laser
  Interventions: Procedure: low-level laser treatment
- Tempormandibular Joint (Experimental): This group with TMD will receive low-level laser treatment in TMJ region - five points around the TMJ.
  Interventions: Procedure: low-level laser treatment
- Withou TMD (No Intervention): This will be a follow up group, with volunteers without TMD.

INTERVENTIONS:
Procedure: low-level laser treatment — A gallium-aluminum-arsenide laser will be employed for the LLLT and placebo treatment. The device will be calibrated with a wavelength of 780 nm, energy density of 25 J/cm2, power of 50 mW and power density of 1.25 W/cm2. Exposure time will be 20 seconds per point, resulting in a total energy of 1 J per point. The spot application method will be used in contact with the skin and with a conventional tip, covering an area of 0.04 cm2.
  Arms: Muscles of mastication; Placebo; TMJ and muscles; Tempormandibular Joint

SUMMARY:
The purpose of this study is to assess the effect of low-level laser on pain, occlusal contacts, mandibular movements and electromyography activity in the masseter and temporal muscles in adolescents with TMD.

DETAILED DESCRIPTION:
A randomized, controlled, double-blind, clinical trial will be carried out. Adolescents aged 15 to 18 years will answer the questionnaire of the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)and a specific clinical exam of RDC/TMD will also be carried out for the diagnosis of temporomandibular disorder (TMD), prior to any intervention. They will also be submitted to electromyographic analysis of the masseter muscles and anterior bundle of the temporal muscles bilaterally for the determination of TMD.

The type of occlusion of those participants will be determined by the clinical examination based on the Angle classification and the occlusal contact points will be recorded using T-Scan III.

Before the intervention, the mandibular range of motion will be assessed by the register of maximum voluntary mouth opening, maximum passive mouth opening and excursion as well as the record pain upon palpation of the masseter and temporal muscles using a visual analog scale.

The volunteers diagnosed with TMD will be divided into four groups and two sessions of LLLT or placebo treatment will be carried out over six weeks. One group will receive low-level laser (LLL) treatment on temporomandibular joint(TMJ) region, one will receive LLL treatment at masseter and temporal muscles, one will receive mixed application of LLL (muscles and TMJ) and the other group will receive placebo treatment.

After the last session of LLL treatment the electromyographic analysis, the record of occlusal contact points, mandibular range of motion and pain upon palpation will be carried out. 30 days following the last session the occlusal contact points, mandibular range of motion and pain upon palpation will be recorded.

Individuals with dentofacial anomalies, incomplete permanent dentition to the 2nd molar, currently undergoing orthodontic or orthopedic treatment of the jaws, currently undergoing psychological treatment or physical therapy and making use of a muscle relaxant, anti-inflammatory agent or bite plate will be excluded from the study.

The data will be submitted to descriptive statistical analysis. The chi-square test and Fisher's exact test will be used for the determination of associations among the categorical variables. The Student's t-test and analysis of variance will be used for the comparison of mean electromyographic signals. Pearson's correlation coefficients will be calculated for the analysis of correlations among the continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 15 to 18 years with diagnosis of TMD and a signed statement of informed consent will be included in the study.

Exclusion Criteria:

* Individuals with dentofacial anomalies, incomplete permanent dentition to the 2nd molar, currently undergoing orthodontic or orthopedic treatment of the jaws, currently undergoing psychological treatment or physical therapy and making use of a muscle relaxant, anti-inflammatory agent or bite plate will be excluded from the study.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyography of masseter and anterior temporal muscles | 6 weeks
  The EMG activity will be read under three conditions: at rest, during chewing (isotonic) and during maximum intercuspation (MI) (isometric). Three readings will be made under each condition, with a three-minute rest interval between readings. The readings in the resting position will be performed, lasting 15 seconds each. The readings under the chewing condition will be performed with the volunteer simulating habitual chewing at a pace determined by a metronome adjusted to 60 beats a minute; lasting 15 seconds each. Three 10-seconds MI readings will be then be performed, with no material placed between the arches, following by three five-second readings during maximum clenching effort (MCE) with a folded layer of Parafilm M® between the molars (bilaterally).

SECONDARY OUTCOMES:
visual analog scale | 10 weeks
  A numeric visual analog scale will be used to record pain upon palpation of the masseter and temporal muscles. It will be applied on the beginning of laser therapy, after 12 sessions of therapy and 30 days following the last session of treatment
mandibular range of motion | 10 weeks
  The volunteer will be instructed to open the mouth as wide as possible. Maximum voluntary mouth opening (distance between upper and lower central incisors) will be recorded with the aid of a digital caliper. The volunteer will then be instructed to exert pressure on the lower teeth with the index and middle finger to obtain maximum passive mouth opening and move the mandible to the right and left for the determination of excursion (distance between upper and lower midpoints).
  These procedures will be carried out at the beginning and end of treatment as well as 30 days following the last session

OTHER OUTCOMES:
occlusal contacts | 10 weeks
  The T-Scan® III will be used for the recording of occlusal contact points. This system is composed of contact sensors connected to a USB port of a computer. Occlusal forces are recorded using a specific software program. The volunteer will be positioned in a chair at 90 degrees such that the Camper plane is parallel to the ground and will be instructed to performed MI.
  It will be recorded before the laser therapy and after the last session fo laser therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Camila HL Godoy, Principal Investigator — University of Nove de Julho; Lara J Motta, Study Chair — University of Nove de Julho; Daniela A Biasotto-Gonzalez, Study Chair — University of Nove de Julho; Fabiano Politti, Study Chair — University of Nove de Julho; Raquel A Mesquita-Ferrari, Study Chair — University of Nove de Julho; Kristianne PS Fernandes, Study Chair — University of Nove de Julho; Sandra K Bussadori, Study Director — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho - Vergueiro, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Carvalho CM, de Lacerda JA, dos Santos Neto FP, Cangussu MC, Marques AM, Pinheiro AL. Wavelength effect in temporomandibular joint pain: a clinical experience. Lasers Med Sci. 2010 Mar;25(2):229-32. doi: 10.1007/s10103-009-0695-y. Epub 2009 Jun 30. PMID 19565312
- [Background] Venezian GC, da Silva MA, Mazzetto RG, Mazzetto MO. Low level laser effects on pain to palpation and electromyographic activity in TMD patients: a double-blind, randomized, placebo-controlled study. Cranio. 2010 Apr;28(2):84-91. doi: 10.1179/crn.2010.012. PMID 20491229
- [Derived] de Godoy CH, Silva PF, de Araujo DS, Motta LJ, Biasotto-Gonzalez DA, Politti F, Mesquita-Ferrari RA, Fernandes KP, Albertini R, Bussadori SK. Evaluation of effect of low-level laser therapy on adolescents with temporomandibular disorder: study protocol for a randomized controlled trial. Trials. 2013 Jul 22;14:229. doi: 10.1186/1745-6215-14-229. PMID 23876095